CLINICAL TRIAL: NCT02613273
Title: CHAMP: A Randomized Controlled Trial of High-intensity Aerobic and Resistance Exercise for Metastatic Prostate Cancer
Acronym: CHAMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 155510; R21CA184605 (NIH); NCI-2017-01928 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2015-11-20; First posted 2015-11-24 (Estimated); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental: Arm 1 (Aerobic Exercise) (Experimental): Arm 1 will engage in a periodized program consisting of 3 aerobic exercise sessions per week comprised of two high-intensity interval training workouts and 1 continuous vigorous intensity workout. A physical assessment, physical function and strengths tests, and questionnaires will be completed at baseline and 3 months.
  Interventions: Behavioral: Experimental: Arm 1 (Aerobic Exercise)
- Experimental: Arm 2 (Resist. Exercise) (Experimental): Arm 2 will engage in a periodized program consisting of 3 resistance exercise sessions per week comprised of various loads and volumes. A physical assessment, physical function and strengths tests, and questionnaires will be completed at baseline and 3 months.
  Interventions: Behavioral: Experimental: Arm 2 (Resist. Exercise)
- No Intervention: Arm 3 (Control) (No Intervention): Arm 3 will follow their usual exercise and lifestyle routine. A physical assessment, physical function and strengths tests, and questionnaires will be completed at baseline and 3 months.

INTERVENTIONS:
Behavioral: Experimental: Arm 1 (Aerobic Exercise) — This periodized program consists of 3 aerobic exercise sessions per week comprised of two high-intensity interval training workouts and 1 continuous vigorous intensity workout.
  Arms: Experimental: Arm 1 (Aerobic Exercise)
Behavioral: Experimental: Arm 2 (Resist. Exercise) — This periodized program consisting of 3 resistance exercise sessions per week comprised of high load/low volume, light load/high volume, and moderate load/moderate volume.
  Arms: Experimental: Arm 2 (Resist. Exercise)

SUMMARY:
This Phase II, open-label, three-arm randomized controlled trial (RCT) will investigate the effects of 12 weeks of aerobic exercise vs. 12 weeks of resistance exercise vs. usual care in men with metastatic castration resistant prostate cancer to determine the safety, feasibility, and tolerance of exercise; quality of life indicators, and a prognostic score.

DETAILED DESCRIPTION:
This is a PI-initiated, randomized clinical trial of 12 weeks of aerobic exercise vs. 12 weeks of resistance exercise vs. usual care among 39 men with metastatic castration resistant prostate cancer. Eligible men will be randomized with equal probability to one of the three regimens. All patients will receive a packet of print material on diet, exercise, and psycho-social support appropriately geared for men with late stage disease at the end of the trial. The aerobic exercise arm (N=13) will receive a 3 day/week remotely-supervised exercise regimen that includes high-intensity interval training and continuous vigorous intensity aerobic exercise training. The resistance exercise arm (N=13) will receive a 3 day/week remotely-supervised resistance exercise regimen incorporating different volumes and loads. Men in the control arm (N=13) will be asked to continue their typical exercise practices for 12 weeks. Subjects will be asked to complete questionnaires, physical function and strength tests, body measurements, and collection of blood specimen at baseline and 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented adenocarcinoma of the prostate with systemic bone or node metastatic disease despite castrate levels of testosterone (<50 ng/dL) due to orchiectomy or luteinising hormone-releasing hormone (LHRH) agonist. Castrate levels of testosterone must be maintained while on study. Men can be enrolled prior to starting abiraterone and/or enzalutamide OR already be receiving treatment with abiraterone and/or enzalutamide.
* On androgen deprivation therapy (ADT) with a Gonadotropin-releasing hormone (GnRH) agonist/antagonist or prior bilateral orchiectomy. All patients will be required to be on ADT throughout the study.
* ≥4 weeks since any major surgery and fully recovered
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Required Initial Laboratory Values:

  * Platelet count ≥ 100,000/microliter (uL)
  * Hepatic and renal dysfunction that would preclude participation in an exercise program, in the opinion of the treating physician
  * Serum testosterone ≤ 50 ng/dL
* Medical clearance to undergo steep ramp test and completion of steep ramp test
* Physician consent to participate in vigorous aerobic or resistance exercise training
* Age ≥18 years

Exclusion Criteria:

* Men with small cell neuroendocrine tumors or features of small cell disease
* Chemotherapy criteria: Metastatic castrate-resistant prostate cancer (CRPC) pre-chemo (metastatic castration-resistant adenocarcinoma prostate cancer, pre-CRPC chemotherapy), which is given for hormone-sensitive prostate cancer, is allowed. Metastatic CRPC post- chemo (metastatic castrate-resistant adenocarcinoma prostate cancer, post-CRPC chemotherapy) is allowed with the treating physician's (oncologist) discretion/approval.
* Poorly controlled hypertension
* Any contraindications to vigorous exercise, including, but not limited to: brain metastases, current congestive heart failure, serious or non-healing wound, and no serious cardiovascular events within 12 months
* Experiences shortness of breath, chest discomfort, or palpitations when performing activities of daily living (can participate with cardiologist clearance)
* Has difficulty climbing a flight of stairs due to physical impairment
* Has been recommended by a doctor to only medically supervised activity
* Has chest pain brought on by physical activity (can participate with cardiologist clearance)
* Has developed chest pain in the past month (can participate with cardiologist clearance)
* Serious or non-healing wound, ulcer, or bone fracture
* Spinal cord compromise or instrumentation due to metastatic disease. Radiation therapy for metastatic disease is allowed.
* Serious or non-healing wound, ulcer, or bone fracture.
* Spinal cord compromise or instrumentation due to metastatic disease. Radiation therapy for metastatic disease is allowed.
* Any peripheral neuropathy ≥grade 3
* Moderate-to-severe bone pain (i.e., National Cancer Institute's Common Terminology Criteria for Adverse Events grade 2-3 bone pain).
* Men participating in vigorous aerobic exercise for 75 minutes or more per week and/or resistance exercise three or more days per week
* Men who do not complete the baseline lifestyle and quality-of-life questionnaires

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2016-07-18 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Number of self-reported adverse events by arm | Up to 4 months
  Adverse events will be assessed at each weekly coach call, at clinic visits during the study, and at the 12-week study visit. They are continuously reported from informed consent until 28 days after the 12-week study visit.
Attendance at 70% or more of exercise sessions. | 3 months
  Study feasibility will be determined by the proportion of participants who complete 70 percent or more of all sessions.
Adherence at 70% or more of the completed exercise sessions. | 3 months
  Study feasibility will be determined by the proportion of participants who completed 70 percent or more of the exercise sessions as or more than prescribed.
Median sessional tolerance | Up to 3 months
  Exercise tolerance will be assessed by participant self-report of a single question at each exercise session using a 10 point Likert scale with a minimum score of 0=intolerable and a maximum score of 10=highly tolerable.
Study acceptability | 3 months
  Proportion of participants who were satisfied or very satisfied with the intervention

SECONDARY OUTCOMES:
Change in scores on the Fatigue visual analog scale (VAS) | 3 months
  Fatigue will be assessed by participant self-report of a single question at each exercise session using a 10 point Likert scale with a minimum score of 0=no fatigue and a maximum score of 10=maximum fatigue.
Change in scores on the Bone pain visual analog scale (VAS) | Up to 3 months
  Bone pain will be assessed by participant self-report of a single question at each exercise session using a 10 point Likert scale with a minimum score of 0=no bone pain and a maximum score of 10=maximum bone pain.
Number of participants reporting use of opiate pain medication | Up to 3 months
  The World Health Organization (WHO) Analgesic Ladder will be used to record the use of pain medication by participants at each visit. The three main principles of the WHO analgesic ladder are: "By the clock, by the mouth, by the ladder". "By the clock" means to maintain freedom from pain, drugs should be given "by the clock" or "around the clock" rather than only "on demand" (i.e. PRN). "By the mouth" means the oral route is usually the preferred route for ease of use in a variety of care settings. "By the ladder" means opiates have been given if pain occurs there should be prompt administration of drugs in the following order: non-opiates (e. g. acetaminophen), as necessary, mild opiates (e. g. codeine), and then strong opiates (e. g. morphine or hydromorphone) until the patient is free of pain. Use of pain medication using the WHO analgesic ladder will be completed at baseline and 3 months.
Change in Scores on the Brief-Pain Inventory Short Form (BPI-SF) | Up to 3 months
  The BPI-SF is a 9-item questionnaire used to assess the severity of pain and the impact of pain on activities of daily living over a recall period of 24 hours. Pain severity is assessed across four sub-scales; 'worst pain', 'least pain', 'average pain' and 'current pain'. A pain score for each subscale is presented separately. Scales are rated on a scale of 0 to 10 (0 = no pain; 10 = pain as bad as one can imagine). A composite score for pain severity is calculated as the mean of the four severity items. Question 9 comprises a 7-item interference scale. Questions assess the level to which pain interferes with general activity, walking, work, mood, enjoyment of life, relations with others and sleep on a scale of 0 to 10 (0 = does not interfere; 10 = completely interferes). Mean interference score will be calculated as an average of the seven subparts of question 9 where at least four of the seven items are completed. Participants will complete the assessment at baseline and 3 months.
Change in objective physical function over time | Up to 3 months
  Participants objective physical function will be assessed using a combination of the the steep ramp (short maximal exercise test that is performed on a cycle ergometer), repeated chair rise, stair climb, and 400 meter (m) walk.
Change in objective physical strength over time | Up to 3 months
  Strength assessments will comprise one repetition maximum (RM)chest press, leg press and seated row. One method will be chosen as the primary method, based on the availability of resistance equipment however, alternative methods will be used, if not appropriate for the patient based on the location of metastasis. The 1-RM is defined as the highest load that can be lifted through full range of movement at one time. Participant suitability to perform each test will be dependent on the site of the metastasis. The decision to either complete or not complete 1 repetition maximum (RM) testing at each site will be decided by the exercise physiologist / therapist performing the test in consultation with the participant's treating physician using an exercise checklist completed by the physician, prior to any testing, which will indicate which exercises to avoid. Any exercise during testing which causes a participant issues will be stopped.
Change in scores on the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) over time | Up to 3 months
  The functional domains measure the quality of life in Physical functioning, Role functioning, Emotional functioning, Cognitive functioning, Social functioning. Scores consists of responses to items with responses ranging from 1="Not at all" to 4="Very Much". The raw score is calculated by estimating the mean of the items that make up each domains with a resulting total range of 1 - 4. These scores are then transformed to standardized scale score, so that scores range from 0 to 100. A high score for the functional domains represents a high level of functioning. Participants will complete the European Organization for Research and Treatment of Cancer (EORTC) QLQ-C30 at baseline and 3 months.
Change in scores on the EuroQol Five-Dimensional Questionnaire (EQ-5D) | Up to 3 months
  EQ-5D is a standardized instrument for measuring generic health status. The health status is measured in terms of five dimensions (5D); mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The respondents self-rate their level of severity for each dimension by selecting one of the following responses: no problems (0), slight problems (1), mild problems (2), moderate problems (3), or severe problems (4) with a particular dimension. Lower scores indicate less issues/problems with that particular health dimension. Participants will complete the EQ-5D at baseline and 3 months.
Change in scores on the Expanded Prostate Cancer Index Composite-26 (EPIC-26) | Up to 3 months
  The EPIC-26 measures the impact of quality of life issues across 5 prostate cancer specific domains: Urinary incontinence, Urinary irritation, Bowel function, Sexual function, and Hormonal function and overall total quality of life. Response options for each EPIC item form a Likert scale, and the raw score of each item is then transformed linearly to a 0-100 scale. Multiple items are combined and then averaged to form the domain scores and total score at each time point also ranging from 0-100, with higher scores representing better health related quality of life (HRQOL). Participants will complete the EPIC-26 at baseline and 3 months.
Change in scores on the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) | Up to 3 months
  The Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) is a 13-item measure that assessing the consequences of fatigue and its impact on participants quality of life. Each item is rated on a 5-point Likert scale ranging from 0 = "Not at all" to 4 = "Very much" with a total score range of 0-52, and higher scores indicating a greater impact of fatigue on . Participants will complete the FACIT-F at baseline and 3 months.
Change in scores on the State-Trait Anxiety Inventory for Adults (STAI) | Up to 3 months
  The Spielberger et. al STAI is a commonly used measure of trait and state anxiety. It can be used in clinical settings to diagnose anxiety and to distinguish it from depressive syndromes. It has 20 items for assessing trait anxiety and 20 for state anxiety for a total of 40 items. State anxiety items include: "I am tense; I am worried" and "I feel calm; I feel secure." Trait anxiety items include: "I worry too much over something that really doesn't matter" and "I am content; I am a steady person." All items are rated on a 4-point scale (e.g., from "1=Almost Never" to 4="Almost Always") with a maximum score range of 40-160 when all 40 items are administered Higher scores indicate greater anxiety. Participants will complete the State Anxiety Inventory at baseline and 3 months.
Change in Scores on the Center for Epidemiological Studies Depression Scale (CESD) | Up to 3 months
  The Center for Epidemiological Studies-Depression (CES-D) is a 20-item measure that asks caregivers to rate how often over the past week they experienced symptoms associated with depression, such as restless sleep, poor appetite, and feeling lonely. Response options range from 0 to 3 for each item (0 = Rarely or None of the Time, 1 = Some or Little of the Time, 2 = Moderately or Much of the time, 3 = Most or Almost All the Time). Scores range from 0 to 60, with high scores indicating greater depressive symptoms. Participants will complete the Center for Epidemiological Studies Depression Scale at baseline and 3 months.
Change in scores on the Pittsburgh Sleep Quality Index (PSQI) over time | Up to 3 months
  The Pittsburgh Sleep Quality Index (PSQI) is a self-rated questionnaire which assesses sleep quality and disturbances over a 1-month time interval. Nineteen individual items generate seven "component" scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The sum of scores for these seven components yields one global score with a possible range of 0-21 points, with lower global scores indicating better sleep overall. Participants will complete the Pittsburgh Sleep Quality Index at baseline and 3 months.
Change in FACT-General (FACT-G) social/family wellbeing domain. | 3 months
  FACT-G SFWB scores range from 0 to 28, with a higher score reflecting better social and familial well-being.

OTHER OUTCOMES:
Number of participants with a change in the Halabi prognostic category over time | 3 months
  An updated prognostic model for patients with prostate cancer was developed by Halabi et. al (2014) which stratifies participants into 3 risk categories: high risk, intermediate risk, or low risk. Risk category is determined by a combination of the following 8 components: albumin levels; alkaline phosphatase levels; Eastern Cooperative Oncology Group Performance Scores; Hemoglobin levels; Lactate dehydrogenase > upper limit of normal, lymph node involvement and prostate-specific antigen (PSA) levels. Participants will be assessed using the Halabi prognostic categorization at baseline and 3 months.
Median Progression-free Survival (PFS) | Up to 2 years
  PFS will be defined as the time from randomization to the date of disease progression + 1 day. Participants who have not progressed at the time of the analysis will be censored on the last date of contact. Participants with no data after randomization will be censored on the day of randomization + 1 day. An intent-to-treat approach will be used to analyze PFS. Data on PFS will be obtained through review of patient medical records at end of study, 1 year, and 2 years. Progression will be determined by the treating physician, and may include any of the following, based on Prostate Cancer Clinical Trials Working Group 3 (PCWG 3) and Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria
Median Overall Survival (OS) | Up to 2 years
  Overall Survival and mortality data will be collected at end of study, one year, and two years through medical records and death records.
Median time to first occurrence of Symptomatic Skeletal-related Events (SSE) | Up to 2 years
  Time to first occurrence of SSE will be defined as the time from randomization to documentation of any of following (whichever occurs first) + 1 day: (1) Use of external beam radiation therapy to relieve bone pain, (2) occurrence of new symptomatic pathological bone fractures that may be vertebral or nonvertebral, asymptomatic compression fractures detected by radiology review only will not be considered a SSE, (3) Spinal cord compression, (4) Change in antineoplastic therapy to treat bone pain, (5) Surgical intervention to treat bone pain. Patients who do not experience a SSE will be censored on the date on which they were last known to be event-free. Adverse events, concomitant medications, concomitant treatment, or survival follow-up case report forms (CRFs) and the participant's medical record will be the source of these findings.

CONTACTS AND LOCATIONS:
Overall Officials: Stacey A Kenfield, ScD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No